CLINICAL TRIAL: NCT04967053
Title: Outcomes of Sleeve Gastrectomy in Obese Patients, Retrospective Study
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Gadelkarim Mohamed, resident doctor, Sohag University
Other Study IDs: Soh-med-21-07-13
Record Dates: First submitted 2021-07-13; First posted 2021-07-19 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; sleeve gastrectomy; bariatric surgery; weight loss
MeSH Terms: conditions — Obesity, Morbid; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: sleeve gastrectomy — Laparoscopic sleeve gastrectomy gives long-standing improvement or resolution of obesity-related conditions and also survival benefit. It is highly cost-effective. Surgical procedures for the treatment of obesity.

SUMMARY:
This study will be a retrospective study in which we will review patients who underwent laparoscopic sleeve gastrectomy at Sohag University Hospital in the period from january 2017 to May 2018.Assessment of outcomes as Effects on weight, Effects on co-morbidities and Post operative complications.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 65 years old
* body mass index ≥ 35 kg/m2 with comorbidities disease or body mass index ≥ 40 kg/m2, with failure of non operative attempts to lose weight
* a minimum 2-year follow-up at our outpatient clinic.

Exclusion Criteria:

* secondary causes of obesity (e.g. endocrine diseases)
* patients unable to participate in medical follow-up;
* associated comorbidities or diseases impacting on weight loss.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: both males and females, age from 18 to 65 yrs complain of obesity with body mass index ≥ 40 kg/m2 or body mass index ≥ 35 kg/m2 with comorbidities diseases.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Effects on weight reported as percentage of excess weight loss | minimum 2-year follow-up
  It is calculated as (initial weight - follow-up weight)/(initial weight - ideal weight corresponding to BMI 25) × 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
participant should be consented for data Sharing